CLINICAL TRIAL: NCT00657709
Title: A Phase 3, Partially Blinded, Randomized, Multi-Center, Controlled Study to Evaluate Immunogenicity, Safety and Lot to Lot Consistency of Novartis Meningococcal B Recombinant Vaccine When Administered With Routine Infant Vaccinations to Healthy Infants
Brief Title: Immunogenicity, Safety and Lot to Lot Consistency of Novartis Meningococcal B Recombinant Vaccine When Administered With Routine Infant Vaccinations to Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P13; EUDRACT 2007-007781-38
Record Dates: First submitted 2008-04-02; First posted 2008-04-14 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-09

CONDITIONS: Serogroup B Meningococcal Meningitis
Keywords: infant; Meningococcal disease; prevention; vaccination
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- rMenB Lot1 (Experimental): Subjects received one injection of rMenB+OMV NZ (Lot 1) at 2, 4, 6 months of age concomitantly with the routinely administered infant vaccines.
  Interventions: Biological: Serogroup B meningococcal Vaccine lot 1 (rMenB Lot 1)
- rMenB Lot2 (Experimental): Subjects received one injection of rMenB+OMV NZ (Lot 2) at 2, 4, 6 months of age concomitantly with the routinely administered infant vaccines.
  Interventions: Biological: Serogroup B meningococcal Vaccine lot 2 (rMenB Lot 2)
- rMenB Lot3 (Experimental): Subjects received one injection of rMenB+OMV NZ (Lot 3) at 2, 4, 6 months of age concomitantly with the routinely administered infant vaccines.
  Interventions: Biological: Serogroup B meningococcal Vaccine lot 3 (rMenB Lot 3)
- Routine (Active Comparator): Subjects received the routinely administered infant vaccines at 2, 4, 6 months of age.
  Interventions: Biological: Infanrix Hexa; Biological: Prevenar
- MenC + Routine (Active Comparator): Subjects received the routinely administered infant vaccines and Men C vaccine at 2, 4 and 6 months of age.
  Interventions: Biological: Infanrix Hexa; Biological: Menjugate; Biological: Prevenar

INTERVENTIONS:
Biological: Serogroup B meningococcal Vaccine lot 1 (rMenB Lot 1) — One dose of rMenB Lot concomitantly with the routinely administered infant vaccines
  Arms: rMenB Lot1
Biological: Serogroup B meningococcal Vaccine lot 2 (rMenB Lot 2) — One dose of rMenB concomitantly with the routinely administered infant vaccines
  Arms: rMenB Lot2
Biological: Serogroup B meningococcal Vaccine lot 3 (rMenB Lot 3) — One dose of rMenB concomitantly with the routinely administered infant vaccines
  Arms: rMenB Lot3
Biological: Infanrix Hexa — Routine vaccination
  Arms: MenC + Routine; Routine
Biological: Menjugate — One dose of the routinely administered infant vaccines + MenC vaccine
  Arms: MenC + Routine
Biological: Prevenar — Routine vaccination
  Arms: MenC + Routine; Routine

SUMMARY:
The proposed study was aimed to assess the immunogenicity, safety, tolerability and lot to lot consistency of 3 lots of Novartis Meningococcal B vaccine when given concomitantly with routine infant vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month old infants (55-89 days, inclusive)

Exclusion Criteria:

* Prior vaccination with routine infant vaccines (Diphtheria, Tetanus, Pertussis, Polio, Haemophilus influenzae type b (Hib), and Pneumococcal antigens)
* Previous ascertained or suspected disease caused by N. meningitidis
* History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component;
* Any serious chronic or progressive disease
* Known or suspected impairment or alteration of the immune system

Ages: 55 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3630 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (66):
- Austria (6):
  - Grässl, Hall in Tirol
  - Häckel, Kirchdorf
  - Prieler, Neufeld A.d. Leitha
  - Maurer, Salzburg
  - Sommer, Vienna
  - Angermayr, Wels
- Czechia (26):
  - Site 27, Boskovice
  - Site 19, Brno
  - Site 22, Chomutov
  - Site11, Červený Kostelec
  - Site 14, Děčín
  - Site 12, Havlíčkův Brod
  - Site 8, Hradec Králové
  - Site 9, Hradec Králové
  - Site 28, Hranice I-mesto
  - Site 13, Humpolec
  - Site 15, Jindřichův Hradec
  - Site 25, Kladno
  - Site 21, Kolín
  - Site 10, Liberec
  - Site 24, Litoměřice
  - Site 17, Ostrava
  - Site 18, Ostrava-Poruba
  - Site 7, Pardubice
  - Site 16, Pilsen
  - Site 2, Prague
  - Site 3, Prague
  - Site 5, Prague
  - Site 6, Prague
  - Site 26, Rumburk
  - Site 23, Ústí nad Labem
  - Site 20, Znojmo
- Finland (15):
  - Site 30, Espoo
  - Site 31, Helsinki
  - Site 32, Helsinki
  - Site 34, Jarvenpaa
  - Site 35, Kokkola
  - Site 45, Kotka
  - Site 46, Kuopio
  - Site 47, Lahti
  - Site 49, Oulu
  - Site 50, Pori
  - Site 51, Seinäjoki
  - Site 52, Tampere
  - Site 53, Turku
  - Site 33, Vantaa
  - Site 48, Vantaa
- Germany (12):
  - Site 99, Detmold
  - Site 92, Espelkamp
  - Site 95, Freising
  - Site 64, Fulda
  - Site 58, Lauffen am Neckar
  - Site 57, Marbach A. N.
  - Site 97, München
  - Site 96, München
  - Site 91, Műnchen
  - Site 81, Porta Westfalica
  - Site 65, Schwieberdingen
  - Site 94, Weilheim
- Italy (7):
  - Dipartimento di Scienze della Salute, Genova
  - Università degli Studi di Messina - Pad. NI - A.O.U. Policlinico G. Martino, Messina
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena Italia, Milan
  - Pediatria dell' Ospedale Sacco, Milan
  - Ospedale Maggiore della Carita'-Clinica Pediatrica, Novara
  - Istituto di Igiene e Medicina Preventiva - Università degli Studi di Sassari, Sassari
  - ASL/TA, Taranto

REFERENCES:
- [Derived] Zafack JG, Bureau A, Skowronski DM, De Serres G. Adverse events following immunisation with four-component meningococcal serogroup B vaccine (4CMenB): interaction with co-administration of routine infant vaccines and risk of recurrence in European randomised controlled trials. BMJ Open. 2019 May 19;9(5):e026953. doi: 10.1136/bmjopen-2018-026953. PMID 31110098
- [Derived] Vesikari T, Esposito S, Prymula R, Ypma E, Kohl I, Toneatto D, Dull P, Kimura A; EU Meningococcal B Infant Vaccine Study group. Immunogenicity and safety of an investigational multicomponent, recombinant, meningococcal serogroup B vaccine (4CMenB) administered concomitantly with routine infant and child vaccinations: results of two randomised trials. Lancet. 2013 Mar 9;381(9869):825-35. doi: 10.1016/S0140-6736(12)61961-8. PMID 23324563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 sites in Finland, 28 sites in the Czech Republic, 13 sites in Germany, 6 sites in Austria, 7 sites in Italy.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- MenC+ Routine: Subjects received the routinely administered infant vaccines and Men C vaccine at 2, 4 and 6 months of age.
Period: Overall Study
Arm/Group | rMenB Lot1 | rMenB Lot2 | rMenB Lot3 | Routine | MenC+ Routine
Started | 833 | 828 | 820 | 659 | 490
Completed | 810 | 795 | 792 | 645 | 457
Not Completed | 23 | 33 | 28 | 14 | 33
Not completed — AE or Death | 7 | 7 | 6 | 7 | 1
Not completed — Withdrawal by Subject | 7 | 15 | 15 | 5 | 9
Not completed — Lost to Follow-up | 9 | 9 | 7 | 1 | 21
Not completed — Protocol Violation | 0 | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rMenB Lot1 | rMenB Lot2 | rMenB Lot3 | Routine | MenC+ Routine | Total
Number analyzed (Participants) | 833 | 828 | 820 | 659 | 490 | 3630
Age, Continuous [Mean (Standard Deviation); unit: Days] | 73.8 (9.5) | 74.1 (9.6) | 73.3 (9.4) | 74.7 (9.3) | 70.6 (9.7) | 73.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 403 | 400 | 416 | 318 | 234 | 1771
  Male | 430 | 428 | 404 | 341 | 256 | 1859

OUTCOME MEASURES:

1. Primary Outcome: The Geometric Mean Human Serum Bactericidal Activity (hSBA) Titers After Three Doses of rMenB+OMV NZ Vaccination
Description: The hSBA antibody titer responses, one month after receiving the third vaccination of rMenB+OMV NZ vaccination, are reported as geometric mean titers (GMTs).
Time Frame: one month after the third vaccination
Population: Analysis was done on Per protocol (PP)population - All subjects who received all the relevant doses of vaccine correctly, and provided evaluable serum samples at the relevant time points, and had no major protocol violation as defined prior to analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB Lot1 | rMenB Lot2 | rMenB Lot3
Number analyzed (Participants) | 386 | 380 | 394
Titers
  44/76-SL strain (Baseline): number analyzed (Participants) | 383 | 379 | 394
  44/76-SL strain (Baseline) | 1.21 [1.14 to 1.29] | 1.19 [1.12 to 1.27] | 1.19 [1.12 to 1.27]
  44/76-SL strain one month after 3rd vaccination: number analyzed (Participants) | 384 | 377 | 388
  44/76-SL strain one month after 3rd vaccination | 87 [80 to 95] | 98 [90 to 106] | 85 [78 to 93]
  5/99 strain (Baseline): number analyzed (Participants) | 385 | 379 | 390
  5/99 strain (Baseline) | 1.21 [1.14 to 1.3] | 1.2 [1.12 to 1.28] | 1.21 [1.13 to 1.29]
  5/99 strain one month after 3rd vaccination: number analyzed (Participants) | 384 | 380 | 388
  5/99 strain one month after 3rd vaccination | 598 [550 to 651] | 681 [626 to 741] | 607 [558 to 661]
  NZ98/254 strain (Baseline) | 1.03 [1 to 1.06] | 1.06 [1.03 to 1.1] | 1.04 [1 to 1.07]
  one month after 3rd vaccination: number analyzed (Participants) | 385 | 378 | 389
  one month after 3rd vaccination | 15 [13 to 17] | 14 [12 to 16] | 15 [14 to 17]
Statistical Analysis 1: Comparison: rMenB Lot1 vs rMenB Lot2; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing rMenB Lot1 to rMenB Lot2 for 44/76-SL strain at one month after the third vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following third vaccination was within this equivalence interval for each of the two co-primary comparisons, rMenB Lot1 and rMenB Lot2 would be equivalent for 44/76-SL strain with respect to the immune response to the vaccine lot; ANOVA; 95% CIs for the GMTs ratios was obtained by exponentiating difference of least square means of log-transformed titers and both the limits of 95% CIs; hSBA GMT ratios = 0.9, 95% CI 2-sided [0.81 to 0.99]
Statistical Analysis 2: Comparison: rMenB Lot1 vs rMenB Lot3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing rMenB Lot1 to rMenB Lot3 for 44/76-SL strain at one month after the third vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following third vaccination was within this equivalence interval for each of the two co-primary comparisons, rMenB Lot1 and rMenB Lot3 would be equivalent for 44/76-SL strain with respect to the immune response to the vaccine lot; ANOVA; [statistical method as in outcome 1, analysis 1]; hSBA GMT ratios = 1.02, 95% CI 2-sided [0.93 to 1.13]
Statistical Analysis 3: Comparison: rMenB Lot2 vs rMenB Lot3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing rMenB Lot2 to rMenB Lot3 for 44/76-SL strain at one month after the third vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following third vaccination was within this equivalence interval for each of the two co-primary comparisons, rMenB Lot2 and rMenB Lot3 would be equivalent for 44/76-SL strain with respect to the immune response to the vaccine lot; ANOVA; [statistical method as in outcome 1, analysis 1]; hSBA GMT ratios = 1.14, 95% CI 2-sided [1.03 to 1.27]
Statistical Analysis 4: Comparison: rMenB Lot1 vs rMenB Lot2; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing rMenB Lot1 to rMenB Lot2 for 5/99 strain at one month after the third vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following third vaccination was within this equivalence interval for each of the two co-primary comparisons, rMenB Lot1 and rMenB Lot2 would be equivalent for 5/99 strain with respect to the immune response to the vaccine lot; ANOVA; [statistical method as in outcome 1, analysis 1]; hSBA GMT ratios = 0.88, 95% CI 2-sided [0.78 to 0.98]
Statistical Analysis 5: Comparison: rMenB Lot1 vs rMenB Lot3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing rMenB Lot1 to rMenB Lot3 for 5/99 strain at one month after the third vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following third vaccination was within this equivalence interval for each of the two co-primary comparisons, rMenB Lot1 and rMenB Lot3 would be equivalent for 5/99 strain with respect to the immune response to the vaccine lot; ANOVA; [statistical method as in outcome 1, analysis 1]; hSBA GMT ratios = 0.99, 95% CI 2-sided [0.88 to 1.1]
Statistical Analysis 6: Comparison: rMenB Lot2 vs rMenB Lot3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing rMenB Lot2 to rMenB Lot3 for 5/99 strain at one month after the third vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following third vaccination was within this equivalence interval for each of the two co-primary comparisons, rMenB Lot2 and rMenB Lot3 would be equivalent for 5/99 strain with respect to the immune response to the vaccine lot; ANOVA; [statistical method as in outcome 1, analysis 1]; hSBA GMT ratios = 1.12, 95% CI 2-sided [1.0 to 1.26]
Statistical Analysis 7: Comparison: rMenB Lot1 vs rMenB Lot2; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing rMenB Lot1 to rMenB Lot2 for NZ98/254 strain at one month after the third vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following third vaccination was within this equivalence interval for each of the two co-primary comparisons, rMenB Lot1 and rMenB Lot2 would be equivalent for for NZ98/254 strain with respect to the immune response to the vaccine lot; ANOVA; [statistical method as in outcome 1, analysis 1]; hSBA GMT ratios = 1.04, 95% CI [0.88 to 1.23]
Statistical Analysis 8: Comparison: rMenB Lot1 vs rMenB Lot3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing rMenB Lot1 to rMenB Lot3 for NZ98/254 strain at one month after the third vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following third vaccination was within this equivalence interval for each of the two co-primary comparisons, rMenB Lot1 and rMenB Lot3 would be equivalent for for NZ98/254 strain with respect to the immune response to the vaccine lot; ANOVA; [statistical method as in outcome 1, analysis 1]; hSBA GMT ratios = 0.96, 95% CI [0.81 to 1.13]
Statistical Analysis 9: Comparison: rMenB Lot2 vs rMenB Lot3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing rMenB Lot2 to rMenB Lot3 for NZ98 /254 strain at one month after the third vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following third vaccination was within this equivalence interval for each of the two co-primary comparisons, rMenB Lot2 and rMenB Lot3 would be equivalent for for NZ98 /254 strain with respect to the immune response to the vaccine lot; ANOVA; [statistical method as in outcome 1, analysis 1]; hSBA GMT ratios = 0.92, 95% CI 2-sided [0.78 to 1.08]

2. Primary Outcome: The Percentages of Subjects With hSBA Titer ≥1:5 After Receiving Three Doses of rMenB+OMV Vaccination (3 Lots Combined)
Description: The immunogenicity was assessed in terms of the percentages of subjects who had received the three doses of rMenB+OMV NZ (3 lots combined) given concomitantly with routine infant vaccinations and percentages of subjects who received only the routine infant vaccinations as measured by hSBA titer ≥1:5 following rMenB+OMV NZ vaccinations one month after the third vaccination is reported.
Time Frame: one month after the third vaccination
Population: Analysis was done on PP population - All subjects who received all the relevant doses of vaccine correctly, and provided evaluable serum samples at the relevant time points, and had no major protocol violation as defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- rMenB All: Subjects received one injection of rMenB+OMV NZ (Lot 1, or Lot 2, or Lot 3) at 2, 4, 6 months of age concomitantly with the routinely administered infant vaccines.
Arm/Group | rMenB All | Routine
Number analyzed (Participants) | 1160 | 121
Percentages of subjects
  44/76-SL strain (Baseline): number analyzed (Participants) | 1156 | 119
  44/76-SL strain (Baseline) | 3 [2 to 4] | 3 [1 to 8]
  44/76-SL strain-1 Month after 3rd vaccination: number analyzed (Participants) | 1149 | 117
  44/76-SL strain-1 Month after 3rd vaccination | 100 [99 to 100] | 3 [1 to 7]
  5/99 strain (Baseline): number analyzed (Participants) | 1154 | 120
  5/99 strain (Baseline) | 4 [3 to 5] | 7 [3 to 13]
  5/99 strain-1 Month after 3rd vaccination: number analyzed (Participants) | 1152 | 116
  5/99 strain-1 Month after 3rd vaccination | 100 [99 to 100] | 2 [0 to 6]
  NZ98/254 strain (Baseline): number analyzed (Participants) | 1160 | 120
  NZ98/254 strain (Baseline) | 1 [1 to 2] | 1 [0.021 to 5]
  1 Month after 3rd vaccination: number analyzed (Participants) | 1152 | 121
  1 Month after 3rd vaccination | 84 [82 to 86] | 2 [0 to 6]

3. Secondary Outcome: The Percentages of Subjects With hSBA Titer ≥1:5 After Receiving Three Doses of rMenB+OMV Vaccination (From 3 Lots)
Description: The immunogenicity was evaluated to assess the consistency of the immune response from three lots of rMenB+OMV NZ in terms of percentage of subjects as measured by hSBA titer ≥1:5 when given to healthy infants at 2, 4, and 6 months of age, at 1 month after the third vaccination.
Time Frame: 1 month after the third vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB Lot1 | rMenB Lot2 | rMenB Lot3 | Routine
Number analyzed (Participants) | 386 | 380 | 394 | 121
Percentages of subjects
  44/76-SL Baseline: number analyzed (Participants) | 383 | 379 | 394 | 119
  44/76-SL Baseline | 4 [2 to 6] | 2 [1 to 4] | 3 [2 to 6] | 3 [1 to 8]
  44/76-SL-1 Month after 3rd vaccination: number analyzed (Participants) | 384 | 377 | 388 | 117
  44/76-SL-1 Month after 3rd vaccination | 100 [99 to 100] | 100 [99 to 100] | 99 [98 to 100] | 3 [1 to 7]
  5/99 Baseline: number analyzed (Participants) | 385 | 379 | 390 | 120
  5/99 Baseline | 3 [2 to 5] | 4 [3 to 7] | 4 [2 to 7] | 7 [3 to 13]
  5/99-1 Month after 3rd vaccination: number analyzed (Participants) | 384 | 380 | 388 | 116
  5/99-1 Month after 3rd vaccination | 100 [99 to 100] | 100 [99 to 100] | 99 [98 to 100] | 2 [0 to 6]
  NZ 98/254 Baseline: number analyzed (Participants) | 386 | 380 | 394 | 120
  NZ 98/254 Baseline | 1 [0 to 2] | 2 [1 to 4] | 1 [0 to 2] | 1 [0.021 to 5]
  1 Month after 3rd vaccination: number analyzed (Participants) | 385 | 378 | 389 | 121
  1 Month after 3rd vaccination | 84 [80 to 88] | 81 [77 to 85] | 85 [81 to 89] | 2 [0 to 6]
Statistical Analysis 1: Comparison: rMenB Lot1 vs rMenB Lot2; The three vaccine lots would be considered equivalent if for each of the three strains and each pair of vaccine lots, the 95% CIs of the differences in the percentage of subjects with hSBA titers ≥ 1:5 at one month after the third vaccination, were entirely within the interval [-10%, 10%]; Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs of the differences in the percentages of subjects at one month following third vaccination was within this equivalence interval for each of the two comparisons, rMenB Lot1 and rMenB Lot2 would be equivalent for 44/76-SL strain; Miettinen and Nurminen; The lot-to-lot differences in these percentages and associated 95% CIs were computed for each pair of rMenB+OMV lots; Vaccines Group Differences = 0, 95% CI 2-sided [-1 to 1]
Statistical Analysis 2: Comparison: rMenB Lot1 vs rMenB Lot3; The three vaccine lots would be considered equivalent if for each of the three strains and each pair of vaccine lots, the 95% CIs of the differences in the percentage of subjects with hSBA titers ≥ 1:5 at 1month after the third dose, were entirely within the interval [-10%, 10%]; Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs of the differences in the percentages of subjects at one month following third vaccination was within this equivalence interval for each of the two comparisons, rMenB Lot1 and rMenB Lot3 would be equivalent for 44/76-SL strain; Miettinen and Nurminen; The lot-to-lot differences in these percentages and associated 95% CIs were computed for each pair of rMenB+OMV lots; Vaccines Group Differences = 1, 95% CI 2-sided [0 to 2]
Statistical Analysis 3: Comparison: rMenB Lot2 vs rMenB Lot3; [analysis description as in outcome 3, analysis 2]; Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs of the differences in the percentages of subjects at one month following third vaccination was within this equivalence interval for each of the two comparisons, rMenB Lot2 and rMenB Lot3 would be equivalent for 44/76-SL strain; Miettinen and Nurminen; The lot-to-lot differences in these percentages and associated 95% CIs were computed for each pair of rMenB+OMV lots; Vaccines Group Differences = 1, 95% CI 2-sided [0 to 2]
Statistical Analysis 4: Comparison: rMenB Lot1 vs rMenB Lot2; [analysis description as in outcome 3, analysis 2]; Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs of the differences in the percentages of subjects at one month following third vaccination was within this equivalence interval for each of the two comparisons, rMenB Lot1 and rMenB Lot2 would be equivalent for 5/99 strain; Miettinen and Nurminen; The lot-to-lot differences in these percentages and associated 95% CIs were computed for each pair of rMenB+OMV lots; Vaccines Group Differences = 0, 95% CI 2-sided [-1 to 1]
Statistical Analysis 5: Comparison: rMenB Lot1 vs rMenB Lot3; [analysis description as in outcome 3, analysis 2]; Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs of the differences in the percentages of subjects at one month following third vaccination was within this equivalence interval for each of the two comparisons, rMenB Lot1 and rMenB Lot3 would be equivalent for 5/99 strain; Miettinen and Nurminen; The lot-to-lot differences in these percentages and associated 95% CIs were computed for each pair of rMenB+OMV lots; Vaccines Group Differences = 1, 95% CI 2-sided [0 to 2]
Statistical Analysis 6: Comparison: rMenB Lot2 vs rMenB Lot3; [analysis description as in outcome 3, analysis 2]; Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs of the differences in the percentages of subjects at one month following third vaccination was within this equivalence interval for each of the two comparisons, rMenB Lot2 and rMenB Lot3 would be equivalent for 5/99 strain; Miettinen and Nurminen; The lot-to-lot differences in these percentages and associated 95% CIs were computed for each pair of rMenB+OMV lots; Vaccines Group Differences = 1, 95% CI 2-sided [0 to 2]
Statistical Analysis 7: Comparison: rMenB Lot1 vs rMenB Lot2; The three vaccine lots would be considered equivalent if for each of the three strains and each pair of vaccine lots, the 95% CIs of the differences in the percentages of subjects with hSBA titers ≥ 1:5 at 1 month after the third dose, were entirely within the interval [-10%, 10%]; Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs of the differences in the percentages of subjects at one month following third vaccination was within this equivalence interval for each of the two comparisons, rMenB Lot1 and rMenB Lot2 would be equivalent for NZ98/254 strain; Miettinen and Nurminen; The lot-to-lot differences in these percentages and associated 95% CIs were computed for each pair of rMenB+OMV lots; Percentage group difference = 3, 95% CI 2-sided [-2 to 8]
Statistical Analysis 8: Comparison: rMenB Lot1 vs rMenB Lot3; The three vaccine lots would be considered equivalent if for each of the three strains and each pair of vaccine lots, the 95% CIs of the differences in the percentage of subjects with hSBA titers ≥ 1:5 at 1 month after the third dise, were entirely within the interval [-10%, 10%]; Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs of the differences in the percentages of subjects at one month following third vaccination was within this equivalence interval for each of the two comparisons, rMenB Lot1 and rMenB Lot3 would be equivalent for NZ 98/254 strain; Miettinen and Nurminen; The lot-to-lot difference in these percentages and associated 95% CIs were computed for each pair of rMenB+OMV lots; Percentage group difference = -1, 95% CI 2-sided [-6 to 4]
Statistical Analysis 9: Comparison: rMenB Lot2 vs rMenB Lot3; The three vaccine lots would be considered equivalent if for each of the three strains and each pair of vaccine lots, the 95% CIs of the differences in the percentage of subjects with hSBA titers ≥ 1:5 at one month after the third dose, were entirely within the interval [-10%, 10%]; Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided (5% CIs of the differences in the percentages of subjects at one month following third vaccination was within this equivalence interval for each of the two comparisons, rMenB Lot2 and rMenB Lot3 would be equivalent for NZ98/254 strain; Miettinen and Nurminen; The lot-to-lot differences in these percentages and associated 95% CIs were computed for each pair of rMenB+OMV lots; Percentage group difference = -4, 95% CI 2-sided [-9 to 1]

4. Secondary Outcome: Geometric Mean Human Serum Bactericidal Activity Titers After the Routine Vaccination Without rMenB OMV NZ
Description: The immunogenicity was assessed in terms of prevalence of meningococcal B antibodies as measured by the hSBA, at baseline and at one month after the third vaccination, in the subjects that received routine infant vaccines without rMenB+OMV NZ.
Time Frame: 1 Month after the third vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- rMenB All: Subjects received one injection of rMenB+OMV NZ (Lot 1, or Lot 2, or Lot 3)at 2, 4, 6 months of age concomitantly with the routinely administered infant vaccines.
Arm/Group | rMenB All | Routine
Number analyzed (Participants) | 1160 | 121
Titers
  44/76 Strain (Baseline): number analyzed (Participants) | 1156 | 119
  44/76 Strain (Baseline) | 1.15 [1.12 to 1.19] | 1.12 [1.04 to 1.22]
  44/76 Strain-1 Month after third vaccination: number analyzed (Participants) | 1149 | 117
  44/76 Strain-1 Month after third vaccination | 91 [87 to 95] | 1.2 [1.1 to 1.31]
  5/99 Strain (Baseline): number analyzed (Participants) | 1154 | 120
  5/99 Strain (Baseline) | 1.18 [1.14 to 1.22] | 1.21 [1.1 to 1.33]
  5/99 Strain-1 Month after third vaccination: number analyzed (Participants) | 1152 | 116
  5/99 Strain-1 Month after third vaccination | 635 [606 to 665] | 1.06 [0.97 to 1.17]
  NZ98/254 (Baseline) | 1.05 [1.03 to 1.07] | 1.01 [0.99 to 1.04]
  1 Month after third vaccination: number analyzed (Participants) | 1152 | 121
  1 Month after third vaccination | 14 [13 to 15] | 1.04 [0.98 to 1.11]

5. Secondary Outcome: Geometric Mean Concentrations After Three Doses of rMenB+OMV NZ Vaccination (Against the 287-953 Antigen)
Description: The immunogenicity was evaluated to characterize the immune response against vaccine antigen 287-953, as measured by ELISA at one month after third vaccination.
Time Frame: 1 month after third vaccination
Population: Analysis was done on PP dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- rMenB All: Subjects received one injection fo rMenB+OMV NZ (Lot1, or Lot 2, or Lot 3) at 2, 4, and 6months of age concomitantly with the routinely administered infant vaccines.
Arm/Group | rMenB Lot1 | rMenB Lot2 | rMenB Lot3 | rMenB All | Routine
Number analyzed (Participants) | 615 | 600 | 611 | 1823 | 113
IU/mL
  Baseline: number analyzed (Participants) | 611 | 596 | 611 | 1818 | 113
  Baseline | 22 [21 to 23] | 22 [21 to 22] | 22 [21 to 23] | 22 [21 to 22] | 21 [20 to 21]
  1 Month after 3rd vaccination: number analyzed (Participants) | 615 | 600 | 608 | 1823 | 113
  1 Month after 3rd vaccination | 3149 [2960 to 3352] | 3484 [3270 to 3712] | 3103 [2915 to 3304] | 3370 [3270 to 3472] | 22 [21 to 23]

6. Secondary Outcome: Geometric Mean Concentrations for Antigens (Pertussis Components) for the Routine Vaccinations
Description: Immunogenicity of the pertussis components (PT, FHA, pertactin) of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 would be considered non-inferior to that of the routine vaccines given alone if the lower limit of the two-sided CI for the ratio of GMCs one month after third vaccination.
Time Frame: 1 month after third vaccination
Population: Analysis was done on Immunogenicity Routine PP (Pertussis Antigens)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | rMenB All | Routine
Number analyzed (Participants) | 241 | 246
IU/mL
  FHA (Baseline) | 9.98 [8.78 to 11] | 9.28 [8.17 to 11]
  1 Month post 3rd vaccination; FHA: number analyzed (Participants) | 239 | 244
  1 Month post 3rd vaccination; FHA | 123 [114 to 133] | 147 [136 to 158]
  Pertactin (Baseline) | 6.3 [5.52 to 7.17] | 5.36 [4.71 to 6.11]
  1 Month post 3rd vaccination; Pertactin: number analyzed (Participants) | 239 | 244
  1 Month post 3rd vaccination; Pertactin | 107 [97 to 119] | 139 [126 to 155]
  PT (Baseline) | 2.82 [2.68 to 2.96] | 2.82 [2.68 to 2.96]
  1 Month post 3rd vaccination; PT: number analyzed (Participants) | 239 | 244
  1 Month post 3rd vaccination; PT | 41 [37 to 44] | 51 [46 to 55]
Statistical Analysis 1: Comparison: rMenB All vs Routine; Immunogenicity of the pertussis components (FHA) of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 would be considered non-inferior to that of routine vaccines given alone if the lower limit of the two-sided CI for the ratio of GMCs one month after the third vaccination is ≥0.67; Test type: Non-Inferiority or Equivalence — GMCs (GMCrMenB+OMV NZ lot1+lot2+lot3+InfanrixHexa / GMCInfanrixHexa); ANOVA; GMCs and 95% CIs were constructed by exponentiating (base 10) the least squares means of the log10-transformed titers and their associated 95% CIs; Geometric group difference = 0.84, 95% CI 2-sided [0.76 to 0.94]
Statistical Analysis 2: Comparison: rMenB All vs Routine; Immunogenicity of the pertussis component (Pertactin) of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 would be considered non-inferior to that of the routine vaccines given alone if the lower limit of the two-sided CI for the ratio of GMCs one month after the third vaccination is ≥0.67; Test type: Non-Inferiority or Equivalence — GMCs (GMCrMenB+OMV NZ lot1+lot2+lot3+InfanrixHexa / GMCInfanrixHexa); ANOVA; GMCs and 95% CIs were constructed by exponentiating (base 10) the least square means of the log10-transformed titers and their associated 95% CIs; Geometric group difference = 0.77, 95% CI 2-sided [0.67 to 0.89]
Statistical Analysis 3: Comparison: rMenB All vs Routine; Immunogenicity of the pertussis components (PT) of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 would be considered non-inferior to that of the routine vaccines given alone if the lower limit of the two-sided CI for the ratio of GMCs one month after the third vaccination is ≥0.67; Test type: Non-Inferiority or Equivalence — GMCs (GMCrMenB+OMV NZ lot1+lot2+lot3+InfanrixHexa / GMCInfanrixHexa); ANOVA; [statistical method as in outcome 6, analysis 1]; Geometric group difference = 0.8, 95% CI 2-sided [0.71 to 0.91]

7. Secondary Outcome: Percentages of Subjects With Antibody Response Against the Routine Antigens
Description: The immunogenicity of routine infant vaccines when given concomitantly with rMenB+OMV NZ at 2, 4, and 6 months of age and of the routine infant vaccines given without rMenB+OMV NZ at 1 month after third vaccination with B pertussis, diptheria and tetanus toxoid, H influenza type b, Hepatitis B antigens was measured by ELISA (Enzyme-linked immunosorbent assay) and for polio type 1, type 2 and type 3 by neutralization test (NT)(>=1:8). Diptheria and Tetanus: primary endpoint ELISA >=0.1 (international unit -IU) IU/mL and the secondary endpoint is ELISA>=1.0 IU/mL.
  HepB (HBV):primary endpoint ELISA >=10 mU/mL. PRP-T: primary endpoint ≥ 0.15 mcg/mL and ≥ 1.00 mcg/mL.PNC >=0.35 mcg/ml
Time Frame: 1 Month after third vaccination
Population: Analysis was done on PP population.
Measure: Number (95% Confidence Interval); unit: Percentages Of Subjects
Arm/Group | rMenB All | Routine
Number analyzed (Participants) | 245 | 252
Percentages Of Subjects
  Anti-DiphtheriaToxin ≥0.1IU/mL(Baseline): number analyzed (Participants) | 241 | 246
  Anti-DiphtheriaToxin ≥0.1IU/mL(Baseline) | 38 [32 to 44] | 38 [32 to 45]
  1 Month post third vaccination;anti-D: number analyzed (Participants) | 239 | 244
  1 Month post third vaccination;anti-D | 100 [98 to 100] | 100 [98 to 100]
  Anti-DiphtheriaToxin ≥1.0 IU/mL(Baseline): number analyzed (Participants) | 241 | 246
  Anti-DiphtheriaToxin ≥1.0 IU/mL(Baseline) | 2 [1 to 5] | 2 [1 to 5]
  1 Month post third vaccination, anti-D≥1.0 IU/mL: number analyzed (Participants) | 239 | 244
  1 Month post third vaccination, anti-D≥1.0 IU/mL | 80 [75 to 85] | 86 [81 to 90]
  Anti-TetanusToxin ≥0.1 IU/mL(Baseline): number analyzed (Participants) | 241 | 246
  Anti-TetanusToxin ≥0.1 IU/mL(Baseline) | 93 [88 to 96] | 95 [91 to 97]
  1 Month post third vaccination;anti-T: number analyzed (Participants) | 239 | 244
  1 Month post third vaccination;anti-T | 100 [98 to 100] | 100 [98 to 100]
  Anti-Tetanus Toxin ≥1.0 IU/mL(Baseline): number analyzed (Participants) | 241 | 246
  Anti-Tetanus Toxin ≥1.0 IU/mL(Baseline) | 24 [18 to 30] | 27 [22 to 33]
  1 Month after third vaccination,anti-T≥1.0 IU/mL: number analyzed (Participants) | 239 | 244
  1 Month after third vaccination,anti-T≥1.0 IU/mL | 91 [86 to 94] | 95 [91 to 97]
  Polio 1 ≥1:8 (Baseline): number analyzed (Participants) | 245 | 246
  Polio 1 ≥1:8 (Baseline) | 75 [69 to 80] | 72 [66 to 77]
  1 Month post third vaccination;Polio 1: number analyzed (Participants) | 243 | 248
  1 Month post third vaccination;Polio 1 | 95 [92 to 98] | 97 [94 to 99]
  Polio 2 (Baseline): number analyzed (Participants) | 245 | 246
  Polio 2 (Baseline) | 68 [62 to 74] | 69 [63 to 74]
  1 Month post third vaccination;Polio 2: number analyzed (Participants) | 243 | 248
  1 Month post third vaccination;Polio 2 | 88 [84 to 92] | 94 [90 to 97]
  Polio 3 (Baseline): number analyzed (Participants) | 245 | 246
  Polio 3 (Baseline) | 48 [41 to 54] | 49 [42 to 55]
  1 Month post third vaccination;Polio 3: number analyzed (Participants) | 243 | 248
  1 Month post third vaccination;Polio 3 | 97 [94 to 99] | 98 [95 to 99]
  HBV ≥10 mIU/mL (Baseline): number analyzed (Participants) | 241 | 248
  HBV ≥10 mIU/mL (Baseline) | 22 [17 to 28] | 15 [10 to 20]
  1 Month post third vaccination;HBV | 98 [95 to 99] | 100 [99 to 100]
  Anti-PRP (HIB) ≥ 0.15 μg/mL(Baseline): number analyzed (Participants) | 241 | 246
  Anti-PRP (HIB) ≥ 0.15 μg/mL(Baseline) | 54 [47 to 60] | 55 [49 to 62]
  1 Month post 3rd vaccination;anti-PRP ≥ 0.15: number analyzed (Participants) | 239 | 244
  1 Month post 3rd vaccination;anti-PRP ≥ 0.15 | 99 [97 to 100] | 100 [98 to 100]
  Anti-PRP (HIB) ≥ 1.0 μg/mL (Baseline): number analyzed (Participants) | 241 | 246
  Anti-PRP (HIB) ≥ 1.0 μg/mL (Baseline) | 12 [9 to 17] | 10 [7 to 15]
  1 Month post third vaccination;anti-PRP ≥ 1.0: number analyzed (Participants) | 239 | 244
  1 Month post third vaccination;anti-PRP ≥ 1.0 | 79 [73 to 84] | 79 [73 to 84]
  PnC4 ≥0.35μg/mL (Baseline): number analyzed (Participants) | 243 | 245
  PnC4 ≥0.35μg/mL (Baseline) | 2 [0 to 4] | 2 [1 to 5]
  1 Month post third vaccination;PnC4: number analyzed (Participants) | 242 | 243
  1 Month post third vaccination;PnC4 | 98 [95 to 99] | 100 [98 to 100]
  PnC 6B ≥0.35μg/mL (Baseline): number analyzed (Participants) | 243 | 245
  PnC 6B ≥0.35μg/mL (Baseline) | 14 [10 to 19] | 16 [12 to 22]
  1 Month post third vaccination;PnC 6B: number analyzed (Participants) | 242 | 243
  1 Month post third vaccination;PnC 6B | 90 [85 to 93] | 88 [83 to 92]
  PnC 9V ≥0.35μg/mL (Baseline): number analyzed (Participants) | 243 | 245
  PnC 9V ≥0.35μg/mL (Baseline) | 4 [2 to 7] | 3 [1 to 6]
  1 Month post third vaccination;PnC 9V: number analyzed (Participants) | 242 | 243
  1 Month post third vaccination;PnC 9V | 100 [98 to 100] | 100 [98 to 100]
  PnC 14 ≥0.35μg/mL (Baseline): number analyzed (Participants) | 243 | 245
  PnC 14 ≥0.35μg/mL (Baseline) | 33 [27 to 39] | 38 [31 to 44]
  1 Month post third vaccination;PnC 14: number analyzed (Participants) | 242 | 243
  1 Month post third vaccination;PnC 14 | 96 [93 to 98] | 97 [94 to 99]
  PnC 18C ≥0.35μg/mL (Baseline): number analyzed (Participants) | 243 | 245
  PnC 18C ≥0.35μg/mL (Baseline) | 10 [7 to 15] | 17 [12 to 22]
  1 Month post third vaccination;PnC 18: number analyzed (Participants) | 242 | 243
  1 Month post third vaccination;PnC 18 | 98 [96 to 100] | 99 [97 to 100]
  PnC 19F ≥0.35μg/mL (Baseline): number analyzed (Participants) | 243 | 245
  PnC 19F ≥0.35μg/mL (Baseline) | 20 [15 to 26] | 21 [16 to 27]
  1 Month post third vaccination;PnC 19: number analyzed (Participants) | 242 | 243
  1 Month post third vaccination;PnC 19 | 96 [93 to 98] | 96 [93 to 98]
  PnC 23F ≥0.35μg/mL (Baseline): number analyzed (Participants) | 243 | 245
  PnC 23F ≥0.35μg/mL (Baseline) | 16 [12 to 21] | 22 [17 to 28]
  1 Month post 3rd vaccination;PnC 23F: number analyzed (Participants) | 242 | 243
  1 Month post 3rd vaccination;PnC 23F | 92 [88 to 95] | 95 [92 to 97]
Statistical Analysis 1: Comparison: rMenB All vs Routine; Immunogenicity of the routine infant vaccines, when given concomitantly with rMenB+OMV NZ at 2, 4, and 6 months of age,would be considered non-inferior to that of routine infant vaccines given alone, for diphtheria toxoids antigen, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response greater than or equal to the cut-off level ≥0.1 IU/mL for that antigen; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = 0, 95% CI 2-sided [-1 to 2]
Statistical Analysis 2: Comparison: rMenB All vs Routine; Immunogenicity of the routine infant vaccines, when given concomitantly with rMenB+OMV NZ at 2, 4, and 6 months of age, would be considered non-inferior to that of routine infant vaccines given alone, for diphtheria toxoids antigen, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response greater than or equal to the cut-off level ≥1.0 IU/mL for that antigen; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = -5, 95% CI 2-sided [-12 to 1]
Statistical Analysis 3: Comparison: rMenB All vs Routine; Immunogenicity of the routine infant vaccines, when given concomitantly with rMenB+OMV NZ at 2, 4, and 6 months of age, would be considered non-inferior to that of routine infant vaccines given alone, for Tetanus toxoids antigen, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response greater than or equal to the cut-off level ≥0.1 IU/mL for that antigen; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 4: Comparison: rMenB All vs Routine; Immunogenicity of the routine infant vaccines, when given concomitantly with rMenB+OMV NZ at 2, 4, and 6 months of age, would be considered non-inferior to that of routine infant vaccines given alone, for Tetanus toxoids antigen, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response greater than or equal to the cut-off level ≥1.0 IU/mL for that antigen; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = -4, 95% CI 2-sided [-9 to 1]
Statistical Analysis 5: Comparison: rMenB All vs Routine; Immunogenicity of the polio type 1 of Diphtheria-Tetanus-Acellular Pertussis, Hepatitis B, Inactivated Poliovirus and Haemophilus influenzae type b (DTPa-HBV-IPV) when given concomitantly with rMenB and Pneumococcal 7-valent conjugate vaccine (PCV7) at 2, 4, and 6 months of age would be considered non-inferior to that of the confidence interval for the difference in the percentage of subjects with NT titers ≥1:8 was greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = -1, 95% CI 2-sided [-5 to 2]
Statistical Analysis 6: Comparison: rMenB All vs Routine; Immunogenicity of the polio type 2 of Diphtheria-Tetanus-Acellular Pertussis, Hepatitis B, Inactivated Poliovirus and Haemophilus influenzae type b (DTPa-HBVIPV) when given concomitantly with rMenB and Pneumococcal 7-valent conjugate vaccine (PCV7) at 2, 4, and 6 months of age would be considered non-inferior to that of the confidence interval for the difference in the percentage of subjects with NT titers ≥1:8 was greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; vaccine group difference = -5, 95% CI 2-sided [-11 to -1]
Statistical Analysis 7: Comparison: rMenB All vs Routine; Immunogenicity of the polio type 3 of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 at 2,4, and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two sided 95% confidence interval for the difference in the percentage of subjects with NT titers ≥1:8 was greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = -1, 95% CI 2-sided [-4 to 2]
Statistical Analysis 8: Comparison: rMenB All vs Routine; Immunogenicity of the hepatitis B surface antigen component of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 vaccine at 2, 4, and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two sided 95% confidence interval for the difference in the percentage of subjects with NT ≥10.0 mIU/ml was greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; percentage group difference = -2, 95% CI 2-sided [-5 to -1]
Statistical Analysis 9: Comparison: rMenB All vs Routine; Immunogenicity of the PRP-Hib component of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 vaccine at 2, 4, and 6 months of age would be considered non-inferiority that of the routine vaccinations given alone, if the lower limit of the two sided 95% confidence interval for the difference in the percentage of subjects with Hib capsular polysaccharide (PRP) antibody response greater than the protective cutoff of ≥0.15 μg/mL was greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; percentage group difference = -1, 95% CI 2-sided [-3 to 1]
Statistical Analysis 10: Comparison: rMenB All vs Routine; Immunogenicity of the PRP-Hib component of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 vaccine at 2, 4, and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two sided 95% confidence interval for the difference in the percentage of subjects with Hib capsular polysaccharide (PRP) antibody response greater than the protective cutoff of ≥1.0 μg/mL was greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; vaccine group difference = 0, 95% CI 2-sided [-7 to 7]
Statistical Analysis 11: Comparison: rMenB All vs Routine; Immunogenicity of the 7 components of PCV7 when given concomitantly with rMenB and DTPa-HBV-IPV at 2, 4 and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two-sided 95% confidence interval for the difference in the percentage of subjects with antibody response greater than the cutoff of ≥0.35 μg/mL was, for the pneumococcal antigen PnC4; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; percentage group difference = -2, 95% CI 2-sided [-4 to 0]
Statistical Analysis 12: Comparison: rMenB All vs Routine; Immunogenicity of the 7 components of PCV7 when given concomitantly with rMenB and DTPa-HBV-IPV at 2, 4, and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response greater than the cutoff of ≥0.35 μg/mL, was, for PnC 6B antigen greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = 2, 95% CI 2-sided [-4 to 8]
Statistical Analysis 13: Comparison: rMenB All vs Routine; Immunogenicity of the 7 components of PCV7 when given concomitantly with rMenB and DTPa_HBV-IPV vaccine at 2, 4, and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two sided 95% CI for the difference in the percentage of subjects with antibody response greater than the cutoff of ≥0.35 μg/mL, was, for PnC 9V, greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = 0, 95% CI 2-sided [-2 to 1]
Statistical Analysis 14: Comparison: rMenB All vs Routine; Immunogenicity of the 7 components of PCV7 vaccine when given concomitantly with rMenB and DTPa-HBV-IPV at 2, 4, and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response greater than the cutoff of ≥0.35 μg/mL, was, for PnC14 antigen, greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = 0, 95% CI 2-sided [-4 to 3]
Statistical Analysis 15: Comparison: rMenB All vs Routine; Immunogenicity of the 7 components of PCV7 when given concomitantly with rMenB and DTPa-HBV-IPV vaccine at 2, 4, and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response greater than the cutoff of ≥0.35 μg/mL, was, for PnC 18C antigen greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = -1, 95% CI 2-sided [-3 to 1]
Statistical Analysis 16: Comparison: rMenB All vs Routine; Immunogenicity of the 7 components of PCV7 when given concomitantly with rMenB and DTPa-HBV-IPV vaccine at 2, 4 and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response greater than the cutoff of ≥0.35 μg/mL, was for PnC 19F antigen, greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = 0, 95% CI 2-sided [-3 to 4]
Statistical Analysis 17: Comparison: rMenB All vs Routine; Immunogenicity of the 7 components of PCV7 when given concomitantly with rMenB and DTPa-HBV-IPV vaccine at 2, 4, and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response greater than the cutoff of ≥0.35 μg/mL, was for PnC 23F antigen, greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = -3, 95% CI 2-sided [-8 to 2]

8. Secondary Outcome: Percentages of Subjects With Fourfold Increase in Antibody Concentrations Against the Routine Antigens
Description: Immunogenicity was assessed in terms of the percentages of subjects with fourfold increase in antibody concentrations against the routine pertussis antigens FHA (Filamentous Hemagglutinin), Pertactin and PT (Pertussis Toxoid).
Time Frame: 5 months
Population: Analysis was done on PP dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | rMenB All | Routine
Number analyzed (Participants) | 238 | 243
Percentages of Subjects
  FHA | 84 [79 to 88] | 87 [82 to 91]
  Pertactin | 79 [73 to 84] | 88 [84 to 92]
  PT | 92 [88 to 95] | 95 [91 to 97]
Statistical Analysis 1: Comparison: rMenB All vs Routine; Immunogenicity of the FHA antigen of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 vaccine at 2, 4 and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects was greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = -3, 95% CI 2-sided [-9 to 4]
Statistical Analysis 2: Comparison: rMenB All vs Routine; Immunogenicity of the Pertactin antigen of DTPa-HBV-IPV when given concomitantly with rMenB and PCV7 at 2, 4 and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects was greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = -9, 95% CI 2-sided [-16 to -3]
Statistical Analysis 3: Comparison: rMenB All vs Routine; Immunogenicity of the PT antigen of DTPa-HBV-IPV vaccine given concomitantly with rMenB and PCV7 vaccine at 2, 4, and 6 months of age would be considered non-inferior to that of the routine vaccinations given alone if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects was greater than -10%; Test type: Non-Inferiority or Equivalence — {PConcomitant Vaccine +rMenB+OMV NZ lot1+lot2+lot3 minus PConcomitant Vaccine}; Miettinen and Nurminen; Percentage group difference = -2, 95% CI 2-sided [-7 to 2]

9. Secondary Outcome: Percentages of Subjects With Fourfold Rise in hSBA Titers After Three Doses of rMenB+OMV NZ Vaccination
Description: Immunogenicity was assessed in terms of the percentages of subjects with fourfold rise in hSBA titers after the three doses of rMenB+OMV NZ (lot 1 or lot 2 or lot 3) vaccination at 2, 4 and 6 months of age.
Time Frame: 1 Month after third vaccination
Population: Analysis was done on PP dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- rMenB Lot1: Subjects received one injection of rMenB+OMV NZ(Lot1) at 2, 4, 6 months of age concomitantly with the routinely administered infant vaccines.
- rMenB Lot3: Subjects received one injection of rMenB+OMV NZ(Lot 3) at 2, 4, 6 months of age concomitantly with the routinely administered infant vaccines.
- rMenB All: Subjects received one injection of rMenB+OMV NZ (Lot 1, or Lot2, or Lot3) at 2, 4, 6 months of age concomitantly with the routinely administered infant vaccines.
Arm/Group | rMenB Lot1 | rMenB Lot2 | rMenB Lot3 | rMenB All | Routine
Number analyzed (Participants) | 370 | 359 | 376 | 1102 | 114
Percentages of Subjects
  44/76-SL: number analyzed (Participants) | 369 | 356 | 373 | 1098 | 111
  44/76-SL | 99 [97 to 100] | 100 [99 to 100] | 98 [97 to 99] | 99 [98 to 100] | 1 [0.023 to 5]
  5/99: number analyzed (Participants) | 370 | 359 | 369 | 1098 | 111
  5/99 | 100 [99 to 100] | 100 [99 to 100] | 99 [98 to 100] | 100 [99 to 100] | 2 [0 to 6]
  NZ98/254: number analyzed (Participants) | 369 | 357 | 376 | 1102 | 114
  NZ98/254 | 70 [66 to 75] | 69 [64 to 74] | 75 [70 to 79] | 71 [69 to 74] | 1 [0.022 to 5]

10. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥1:8
Description: Immunogenicity was assessed in terms of the percentages of subjects achieving hSBA titers ≥1:8 at one month after third vaccination with rMenB (lot 1 or lot 2 or lot 3) against the three vaccine strains.
Time Frame: 1 month after third vaccination
Population: Analysis was done on PP population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- rMenB Lot2: Subjects received one injection of rMenB+OMV NZ(Lot 2) at 2, 4, 6 months of age concomitantly with the routinely administered infant vaccines.
Arm/Group | rMenB Lot1 | rMenB Lot2 | rMenB Lot3 | rMenB All | Routine
Number analyzed (Participants) | 386 | 379 | 394 | 1156 | 119
Percentages of subjects
  44/76-SL (Baseline): number analyzed (Participants) | 383 | 379 | 394 | 1156 | 119
  44/76-SL (Baseline) | 2 [1 to 4] | 2 [1 to 3] | 2 [1 to 4] | 2 [1 to 3] | 2 [0 to 6]
  1 Month after 3rd vaccination-44/76-SL: number analyzed (Participants) | 384 | 377 | 388 | 1149 | 117
  1 Month after 3rd vaccination-44/76-SL | 100 [99 to 100] | 100 [99 to 100] | 99 [98 to 100] | 100 [99 to 100] | 1 [0.022 to 5]
  5/99 (Baseline): number analyzed (Participants) | 385 | 379 | 390 | 1154 | 119
  5/99 (Baseline) | 3 [1 to 5] | 3 [1 to 5] | 2 [1 to 4] | 3 [2 to 4] | 2 [0 to 6]
  1 Month after 3rd vaccination-5/99: number analyzed (Participants) | 384 | 379 | 388 | 1152 | 116
  1 Month after 3rd vaccination-5/99 | 100 [99 to 100] | 100 [99 to 100] | 99 [98 to 100] | 100 [99 to 100] | 2 [0 to 6]
  NZ98/254 (Baseline) | 1 [0.063 to 2] | 1 [0 to 3] | 0 [0 to 1] | 1 [0 to 1] | 0 [0 to 3]
  1 Month after 3rd vaccination: number analyzed (Participants) | 385 | 378 | 389 | 1152 | 119
  1 Month after 3rd vaccination | 70 [66 to 75] | 70 [65 to 74] | 75 [70 to 79] | 72 [69 to 74] | 1 [0.021 to 5]

11. Secondary Outcome: Number of Subjects Reporting Solicited Adverse Events After Receiving Three Doses of rMenB+OMV NZ Vaccine
Description: The safety and tolerability of three doses of rMenB+OMV NZ when given concomitantly with routine infant vaccines at 2, 4 and 6 months of age was assessed by the number of subjects reporting solicited local and systemic adverse events.
Time Frame: upto 7 days after any vaccination
Population: The analysis was done on safety subset population - all subjects enrolled who received study vaccination and provided post-baseline safety data.
Measure: Number; unit: Participants
Groups:
- MenC+Routine: Subjects received the routinely administered infant vaccines and MenC vaccine at 2, 4 and 6 months of age.
Arm/Group | rMenB All | MenC+Routine
Number analyzed (Participants) | 2479 | 490
Participants
  Any Local | 2388 | 443
  Injection site tenderness | 2147 | 266
  Injection site erythema | 2049 | 261
  Injection site induration | 1908 | 227
  Injection site swelling | 1174 | 84
  Any Systemic | 2450 | 459
  Change in Eating Habits | 1787 | 257
  Sleepiness | 2159 | 353
  Vomiting | 662 | 116
  Diarrhea | 1086 | 164
  Irritability | 2296 | 370
  Unusual Crying | 2109 | 352
  Rash | 318 | 43
  Fever >= 38.5C | 1912 | 228
  Others | 2302 | 325
  Medical Attend. Fever | 57 | 16
  Analg. Antipyretic Med.Used | 2302 | 325
  Antipyretic Med.Used | 2240 | 314

ADVERSE EVENTS:
Time Frame: All serious adverse events and medically attended adverse events are collected from Day 8 after each vaccination to next vaccination or to 30 days after the last vaccination.
Description: Of a total of 3630 enrolled subjects, 3629 received at least one vaccination and were included in the safety analysis.
Arm/Group | rMenB Lot1 | rMenB Lot2 | rMenB Lot3 | Routine | MenC+Routine
Serious Adverse Events (participants affected / at risk) | 70/832 | 80/828 | 60/820 | 51/659 | 28/490
Other Adverse Events (participants affected / at risk) | 827/832 | 825/828 | 817/820 | 652/659 | 482/490
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB Lot1 (N=832) | rMenB Lot2 (N=828) | rMenB Lot3 (N=820) | Routine (N=659) | MenC+Routine (N=490)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cerebral Palsy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Congenital Coronary Artery Malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Faciodigitogenital Dysplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Gnathoschisis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Microcephaly (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Thalassaemia Beta (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 1 | 0 | 0 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 0
Enteritis (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Infantile Colic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intusscusception (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Irritability (General disorders) | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 3 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Milk allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bacterial Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 4 | 2 | 5 | 0 | 2
Bronchitis (Infections and infestations) | 6 | 12 | 7 | 11 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 4 | 1 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Exanthema Subitum (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Febrile Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 12 | 7 | 12 | 7 | 2
Gastroenteritis Adenovirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 3 | 4 | 1 | 1 | 2
Gastroenteritis Salmonella (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 7 | 4 | 3 | 3 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 2 | 0
Otitis media (Infections and infestations) | 3 | 2 | 6 | 3 | 0
Otitis media acute (Infections and infestations) | 2 | 1 | 0 | 1 | 0
Pertussis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 4 | 3 | 2 | 1
Pseudocroup (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 3 | 6 | 2 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 3 | 3 | 2 | 0
Respiratory syncytial virus (Infections and infestations) | 1 | 0 | 0 | 2 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
H1N1 Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tonsilitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 3
Varicella (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Accidental exposure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 2 | 0
Foregin body trauma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Feeding disorder or infancy or early childhood (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Premature closure of cranial sutures (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 2 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 1 | 1 | 3 | 0 | 0
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Infantile spasms (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Breath Holding (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Decreased activity (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Eczema Nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Labial frenectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Tendon operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Kawasaki's disease (Vascular disorders) | 1 | 1 | 1 | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rMenB Lot1 (N=832) | rMenB Lot2 (N=828) | rMenB Lot3 (N=820) | Routine (N=659) | MenC+Routine (N=490)
Cough (Respiratory, thoracic and mediastinal disorders) | 59 (66) | 58 (66) | 60 (69) | 43 (48) | 40 (51)
Somnolence (Nervous system disorders) | 714 (1657) | 729 (1684) | 716 (1624) | 476 (914) | 353 (711)
Crying (General disorders) | 714 (1740) | 711 (1750) | 685 (1693) | 424 (822) | 352 (752)
Injection site erythema (General disorders) | 729 (4171) | 733 (4135) | 704 (4034) | 497 (1792) | 385 (1788)
Injection site induration (General disorders) | 692 (4024) | 680 (3915) | 664 (3926) | 452 (1741) | 390 (1761)
Injection site pain (General disorders) | 736 (4472) | 736 (4497) | 728 (4541) | 415 (1364) | 358 (1615)
Injection site swelling (General disorders) | 440 (1683) | 466 (1688) | 436 (1743) | 254 (653) | 184 (519)
Pyrexia (General disorders) | 656 (1344) | 646 (1338) | 643 (1332) | 319 (493) | 248 (425)
Vaccination site induration (General disorders) | 42 (76) | 30 (60) | 38 (74) | 4 (5) | 51 (105)
Eating disorder (Psychiatric disorders) | 588 (1152) | 603 (1223) | 596 (1211) | 329 (580) | 257 (492)
Irritability (Psychiatric disorders) | 769 (2181) | 761 (2168) | 766 (2183) | 544 (1339) | 370 (877)
Diarrhoea (Gastrointestinal disorders) | 370 (607) | 380 (632) | 368 (624) | 225 (358) | 168 (286)
Vomiting (Gastrointestinal disorders) | 217 (315) | 234 (329) | 216 (317) | 108 (149) | 120 (178)
Rash (Skin and subcutaneous tissue disorders) | 121 (180) | 119 (168) | 110 (147) | 88 (116) | 50 (79)
Bronchitis (Infections and infestations) | 102 (129) | 98 (132) | 94 (123) | 97 (125) | 59 (80)
Conjunctivitis (Infections and infestations) | 74 (91) | 80 (100) | 77 (91) | 60 (66) | 16 (19)
Ear infection (Infections and infestations) | 86 (119) | 70 (106) | 57 (85) | 59 (91) | 26 (38)
Exanthema subitum (Infections and infestations) | 46 (46) | 47 (47) | 46 (46) | 38 (38) | 21 (21)
Gastroenteritis (Infections and infestations) | 34 (34) | 47 (51) | 38 (41) | 25 (25) | 14 (15)
Nasopharyngitis (Infections and infestations) | 78 (97) | 79 (108) | 81 (106) | 73 (107) | 12 (12)
Otitis media (Infections and infestations) | 152 (256) | 145 (267) | 156 (284) | 124 (229) | 28 (38)
Rhinitis (Infections and infestations) | 78 (90) | 99 (120) | 58 (66) | 63 (84) | 30 (33)
Upper respiratory tract infection (Infections and infestations) | 142 (190) | 126 (172) | 133 (175) | 94 (124) | 47 (59)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days